CLINICAL TRIAL: NCT04744259
Title: Behavioural Activation (BeatIt) for Depression in Adults With Severe Intellectual Disabilities. A Feasibility Randomised Controlled Study of BeatIt Versus Treatment as Usual
Brief Title: BEAT-IT: Behavioural Activation and Severe Learning Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); Lancaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN18MH490
Record Dates: First submitted 2019-03-05; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Depression
Keywords: Intellectual Disability
MeSH Terms: conditions — Depression; Intellectual Disability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioural activation (Experimental): The treatment is designed to be delivered to individuals alongside a carer who provides regular support to them. It is a structured, time limited, manualised psychological therapy, developed to treat those with an intellectual disability and depressive symptoms.
  Interventions: Behavioral: Behavioural Activation
- Treatment as usual (No Intervention): This will include the existing treatments available in NHS and social care for adults with intellectual disability with depression, including anti-depressants, mood stabilizers, and any available psychological interventions. Additionally, for all those in the study, we will provide their General Practitioner with a summary of the NICE guidelines on treatment of depression for adults with intellectual disabilities.

INTERVENTIONS:
Behavioral: Behavioural Activation — A psychological intervention which aims to increase activity and reduce depressive symptoms.
  Arms: Behavioural activation

SUMMARY:
Depression is common, but no psychological interventions have been tested to see if they work for adults with severe intellectual disabilities. The research team recently successfully completed a full-scale trial of a psychological intervention, BeatIt, for depressed adults with mild/moderate intellectual disabilities. The aim of this study is to comprehensively evaluate the feasibility of modifying BeatIt for depressed adults with severe intellectual disabilities, collecting the information needed on likely recruitment, measures, and waiting list control arm options, to design a full-scale study.

ELIGIBILITY:
Inclusion Criteria:

* Severe/profound intellectual disabilities
* 18 years old and over
* Clinically significant unipolar depression
* Has a family member or paid carer who has supported them for a minimum of 6 months to complete the screening and baseline visits OR is able to obtain information for the previous 4 months prior to randomisation. The carer, or another named individual, should be available for weekly-fortnightly treatment sessions with the practitioner, and should currently provide a minimum of 10 hours support per week to the participant.

Exclusion Criteria:

* Suicidal
* Mild/moderate intellectual disabilities
* Factors that prevent the person from interacting with the carer and therapist or retaining information from the therapy (e.g. late stage dementia, significant agitation, withdrawal arising from psychosis)
* Does not consent to her/his GP being contacted about their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the Mood, Interest and Pleasure Questionnaire (MIPQ) at 24 weeks | Baseline and week 24
  A measure of the individuals mood and engagement in activities. The score range for each sub-scale is 0 - 24.
  Total score range is 0 - 48. Lower scores indicate lower mood and lower levels of interest and pleasure (within the last 2 week)
Change from baseline on Intellectual Disabilities Depression Scale (IDDS) at 24 weeks | Baseline and week 24
  This is a 38-item behavioural checklist derived from DSM-III-R criteria, designed to measure the frequency of identified depressive behaviours within a four-week period. Each item is scored on a 7-point Likert scale from 0 (never) to 6 (always). All scores are summed to provide a total score, ranging from 0 to 228. Higher scores indicate a higher frequency of depressive symptoms.

SECONDARY OUTCOMES:
Change from baseline on the Anxiety, Depression and Mood Scale at 24 weeks | Baseline and week 24
  This scale has been shown to be a reliable and valid measure of anxiety in adults with severe/profound intellectual disabilities. The 7 item 'generalised anxiety' sub-scale was used.
  Items are rated on a four-point Likert scale for frequency from 0 (never) to 3 (always) and for severity 0 (not a problem) to 3 (severe problem). Items are based on informants' observations in the last 2 weeks. Scores are summed. The possible score range for frequency of anxiety symptoms is 0-21, total score range for severity of anxiety symptoms is 0 - 21 and total score is 0 - 42. Higher scores indicate a higher frequency of anxiety symptoms and higher severity of anxiety symptoms.
Change from baseline on the Modified Index of Community Involvement (ICI) at 24 weeks | Baseline and week 24
  This scale provides a measure of participation in social and community-based activities during the previous 4 weeks. This is a 16-item scale, measuring participation in social activities (5 items), community activities (10 items) and going on holiday (1 item).
  The informant is asked to rate whether the participant has participated in any of these events in the last month (12 months for the item 'been on holiday'), and if so, how many times (once through to five times or more). All items are rated on a 6-point Likert scale (0 = not participated, 5 = participated 5x or more). All scores are summed. The possible score range for the social activities sub-scale is 0-25, the possible score range for the community activities subscale is 0-50 and the total scale score range is 0-80. Higher scores indicate a higher frequency of engagement in social and community activities.
Change from baseline on the Modified Index of Domestic Participation at 24 weeks | Baseline and week 24
  This scale measures participation in 13 household tasks during the previous 4 weeks. All items are rated on a three-point Likert scale (0 - no participation, 1 - participation with help, 2 - independent participation). Scores are summed, with a possible score range of 0 - 26. Higher scores indicate higher levels of independent participation in domestic tasks.
Change from baseline on the Emotional Difficulties self-efficacy scale at 24 weeks | Baseline and week 24
  This is a 10-item scale which measures the carer's confidence in supporting the person when they are feeling down. All item are scored on a 9-point Likert scale, where 0 indicates 'not at all confident' and 8 indicates 'extremely confident'. All scores are summed with a possible score range of 0 - 80. Higher scores indicate a higher level of self-confidence in supporting someone when they are feeling down.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Jahoda, PhD, Principal Investigator — Professor of Learning Disabilities
Locations (1):
- Institute of Health and Wellbeing, University of Glasgow, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No